CLINICAL TRIAL: NCT05874050
Title: The Effect of Arterial Pressure on Surgical Hemostasis During Elective Supratentorial Neurosurgery: a Prospective Observational Study.
Brief Title: Arterial Pressure and Surgical Hemostasis in Elective Neurosurgery.
Acronym: HemoStopArt
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fondazione I.R.C.C.S. Istituto Neurologico Carlo Besta (Other)
Responsible Party: Sponsor
Other Study IDs: Ria2022_01
Record Dates: First submitted 2023-05-16; First posted 2023-05-24 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: Neurosurgery; Intracranial Hemorrhages; Supratentorial Brain Tumor; Blood Pressure
MeSH Terms: conditions — Intracranial Hemorrhages

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The objective of this observational study is to examine the impact of augmented arterial pressure during the hemostatic phase of elective supratentorial neurosurgery. The primary inquiries it seeks to address are as follows:

1. Does an increase in systolic arterial pressure prompt a hemostatic maneuver by the neurosurgeon, and does the concomitant mean arterial pressure value influence the frequency of such interventions?
2. How often do postoperative intracranial hemorrhages occur, and how severe are they in relation to the achieved mean arterial pressure value?

Participants will be enrolled during the preoperative evaluation, where their arterial pressure values, medical histories, and medication statuses will be recorded. Throughout the induction and maintenance of anesthesia, we will monitor their blood pressure values and document any instances of hypotension or hypertension. During the hemostatic phase, we will elevate the arterial pressure using noradrenaline by up to 10 mmHg above the recorded pressure measured at the inpatient clinic. Subsequently, we will inquire whether the neurosurgeon had to employ any additional hemostatic maneuvers following the increase in arterial pressure. The arterial pressure values will be recorded at the end of the surgery, and the first postoperative CT scan will be examined to identify any cases of intracranial hemorrhage.

DETAILED DESCRIPTION:
During surgery to remove intracranial tumors, a patient's blood pressure is kept moderately low to facilitate the procedure. Subsequently, a surgical phase of hemostasis is performed. At this stage, the standard clinical practice requires the anesthesiologist to raise blood pressure to challenge the surgical hemostasis. Although this practice may be considered ubiquitous, it is not currently described in neuroanesthesia texts, and no studies are available that report the effect of this maneuver, either in terms of the optimal level of pressure elevation or in terms of the greater efficacy of a target of systolic arterial pressure (SAP) rather than mean arterial pressure (MAP). The most frequently sought increase in everyday clinical practice is about 10 mmHg higher than the first SAP measured in the patient's operating room. Because of the different profiles of brain autoregulation (Smith, 2015) and individual cardiovascular profiles, anticipatory and context anxiety accompanying the time of surgery, in line with the literature, the present study prefers to select the blood pressure value measured on the ward at the time of admission as the reference (Ackland et al., 2019; Ard & Kendale, 2016). The study aims first to observe the effects on the operative field of this increase.

* Primary objective: To verify how frequently the SAP-increasing maneuver prompts the Neurosurgeon to perform a hemostatic maneuver on the surgical field and to evaluate whether the concomitant MAP value reached affects this frequency.
* Secondary objective: To quantify the frequency and severity of any postoperative intracranial hemorrhage in relation to the achieved MAP value.

There are no pharmacological strategies to increase SAP and MAP selectively. However, it can be estimated that the increase mentioned above in SAP, achieved in our institute with an intravenous norepinephrine infusion, is not accompanied by a parallel increase in MAP in about 50 percent of cases (unpublished data).

ELIGIBILITY:
Inclusion Criteria:

* All consecutive adult patients scheduled to undergo elective supratentorial neurosurgical surgery.

Exclusion criteria:

* Urgent or emergent surgery
* Neurovascular surgery
* Subtentorial surgery
* Trans nasal approaches
* Back surgery
* Acute or chronic kidney injury as defined according to the Kidney Disease: Improving Global Outcomes (KDIGO) guidelines (Kellum & Lameire, 2013; Stevens & Levin, 2013)
* Coagulation derangement (platelet count < 100*10^9/L, international normalized ratio (INR) or activated partial thromboplastin time (aPTT) > 1.5 times the normal laboratory range) or anticoagulant/antiplatelet treatment without appropriate withhold intervals, as per existing guidelines
* Preoperative severe hemodynamic instability, according to the judgment of the attending physician
* Age < 18 years
* Pregnancy or breastfeeding
* Absence of informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive adult patients scheduled to undergo elective supratentorial neurosurgical surgery.
Sampling Method: Non-Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2022-11-11 (Actual); Primary Completion 2024-02-27 (Estimated); Study Completion 2024-02-27 (Estimated)

PRIMARY OUTCOMES:
Frequency of need for hemostatic maneuver in the neurosurgical field | During surgery
  We document the frequency with which the primary operators indicate the need for additional maneuvers once the target systolic arterial pressure (SAP) exceeds a 10 mmHg increase from the baseline relative to the achieved mean arterial pressure (MAP) value.
Number of postoperative neurosurgical site hemorrhage requiring treatment | In the 24 hrs after surgery
  In relation to the MAP value achieved, we register the number of times the presence of a neurosurgical site hemorrhage calls for a novel surgical treatment or significant therapy adjustments.

CONTACTS AND LOCATIONS:
Overall Officials: Marco Fabio Gemma, Dr, Principal Investigator — Fondazione IRCCS Istituto Neurologico Carlo Besta Milan, Italy
Locations (1):
- Fondazione IRCCS Istituto Neurologico C. Besta, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided